CLINICAL TRIAL: NCT01918007
Title: Adenotonsillectomy for Obstructive Sleep-Disordered Breathing in Childhood:The Chania Community Oximetry-Based Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chania General Hospital "St. George" (Other)
Collaborators: Aghia Sophia Children's Hospital of Athens (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CHANIA-ENT-01
Record Dates: First submitted 2013-07-26; First posted 2013-08-07 (Estimated); Results first posted 2023-11-13 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2020-08

CONDITIONS: Sleep Disordered Breathing; Obstructive Sleep Apnea; Snoring; Obstructive Sleep Disordered Breathing
Keywords: Apnea; Sleep Apnea Syndromes; Snoring; Sleep Apnea, Obstructive; Respiration Disorders; Respiratory Tract Diseases; Signs and Symptoms, Respiratory Signs and Symptoms; Sleep Disorders, Intrinsic; Dyssomnias; Sleep Disorders; Respiratory Sounds
MeSH Terms: conditions — Sleep Apnea Syndromes; Sleep Apnea, Obstructive; Snoring; Apnea; Respiration Disorders; Respiratory Tract Diseases; Signs and Symptoms, Respiratory; Sleep Disorders, Intrinsic; Dyssomnias; Sleep Wake Disorders; Respiratory Sounds | interventions — Adenoidectomy

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- AT (adenotonsillectomy) Group (Active Comparator): AT (adenotonsillectomy) immediately after the baseline study evaluation
  Interventions: Procedure: Adenotonsillectomy (AT)
- Control Group (No Intervention): No AT (adenotonsillectomy) for 3 months after the baseline study evaluation

INTERVENTIONS:
Procedure: Adenotonsillectomy (AT) — Standard surgical intervention for treatment of obstructive sleep-disordered (SDB).
  Other Names: Removal of adenoids and tonsils
  Arms: AT (adenotonsillectomy) Group

SUMMARY:
Obstructive sleep-disordered breathing (SDB) in childhood is a disorder of breathing during sleep characterized by intermittent upper airway obstruction. Snoring, labored breathing and apneas reported by the parents are the most frequent symptoms.Obstructive SDB can result from many different abnormalities including large adenoids and tonsils or obesity.

Intermittent upper airway obstruction during sleep is accompanied by low oxygen or high carbon dioxide in the blood and arousals from sleep. If obstructive SDB is not treated, complications may develop such as: i) enuresis; ii) delay in somatic growth rate; iii) central nervous system morbidity (e.g. hyperactivity and learning difficulties); and iv) elevated blood pressure.

Overnight polysomnography (PSG) is considered the gold-standard method for defining severity of obstructive SDB and subgroups of children with snoring who should be treated. However, PSG is a labor-intensive, time-consuming and expensive diagnostic method, which is not available in many community settings. Thus, there is an urgent need for developing easy-to-use and low-cost diagnostic methods which can be used to determine severity of obstructive SDB and define subgroups of children with snoring and large adenoids and tonsils who will benefit from adenotonsillectomy (AT).

Pulse oximetry is a widely available, non-invasive method which allows continuous monitoring of oxygen transport by hemoglobin. Episodes of upper airway obstruction are frequently accompanied by reductions in the hemoglobin oxygen transport (oxygen desaturation of hemoglobin).The hypothesis of this research project is that subgroups of children with snoring and adenotonsillar hypertrophy and certain abnormalities in oxygenation detected by nocturnal pulse oximetry will benefit from AT in a community setting.

DETAILED DESCRIPTION:
Time in the waiting list for undergoing AT at the Department of Otorhinolaryngology, Chania General Hospital "St. George" is approximately 3 months. In the present study, children will be recruited and randomized in the Active Comparator (AT group) or in the Control Group (No AT group) at the time of the initial clinic visit, if they fulfill the Inclusion Criteria and their parents consent to participation in the study.

Children in the AT group will undergo the baseline study evaluation at the end of the 3-month waiting time and thus immediately prior to AT. They will also undergo the follow-up study evaluation at 3 months postoperatively.

Children in the Control group will undergo their baseline study evaluation at the time of entering the surgical waiting list. They will undergo the follow-up study evaluation 3 months later, immediately prior to AT.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with obstructive SDB (snoring >3 nights/week over the last 6 months)
* Tonsillar size >2 [Brodsky 1989]
* Considered as an AT candidate during the clinic visit by ear, nose and throat (ENT) surgeon

Exclusion Criteria:

* Recurrent tonsillitis defined as at least 3 episodes in each of the last 3 years or at least 5 episodes in each of the last 2 years or at least 7 episodes in the past year.
* Apparent craniofacial anomalies (e.g. Crouzon syndrome or Pierre-Robin sequence)
* Obstructive breathing while awake or any other clinical signs that merit prompt AT as recommended by the treating ENT physician.
* History of clinically important cardiovascular disease or cardiac arrhythmia.
* History of: sickle cell disease; symptomatic asthma; epilepsy; use of sedative medication
* History of: genetic disorders; neurological or neuromuscular disorders
* Use of: systemic or intranasal corticosteroids; montelukast

Footnote

Brodsky score Upon inspection of the oropharynx

* grade 1 indicates that the tonsils are hidden in the pillars
* grade 2 indicates that the tonsils are beyond the anterior pillar and occupy between 25 and 50% of the pharyngeal space
* grade 3 indicates that the tonsils are beyond the pillars but not to the middle and occupy >50% and up to 75% of the pharyngeal space
* grade 4 indicates that the tonsils occupy >75% of the pharyngeal space

Ages: 4 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 186 (Actual)
Dates: Start 2013-06; Primary Completion 2016-04 (Actual); Study Completion 2016-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chariton E. Papadakis, MD, Study Director — Chania General Hospital "St. George"; Athanasios G. Kaditis, MD, Study Chair — Aghia Sophia Children's Hospital of Athens; Theognosia S. Chimona, MD, Principal Investigator — Chania General Hospital "St. George"; Panagiota N. Asimakopoulou, MD, Principal Investigator — Chania General Hospital "St. George"; Efklidis Proimos, MD, Principal Investigator — Chania General Hospital "St. George"; Konstantinos Chaidas, MD, Principal Investigator — Aghia Sophia Children's Hospital of Athens; Alexandra Klimentopoulou, MD, Principal Investigator — Aghia Sophia Children's Hospital of Athens
Locations (2):
- Greece (2):
  - Aghia Sophia Children's Hospital of Athens, Athens
  - Chania General Hospital "St. George", Chania

REFERENCES:
- [Background] Nixon GM, Kermack AS, Davis GM, Manoukian JJ, Brown KA, Brouillette RT. Planning adenotonsillectomy in children with obstructive sleep apnea: the role of overnight oximetry. Pediatrics. 2004 Jan;113(1 Pt 1):e19-25. doi: 10.1542/peds.113.1.e19. PMID 14702490
- [Background] Saito H, Araki K, Ozawa H, Mizutari K, Inagaki K, Habu N, Yamashita T, Fujii R, Miyazaki S, Ogawa K. Pulse-oximetery is useful in determining the indications for adeno-tonsillectomy in pediatric sleep-disordered breathing. Int J Pediatr Otorhinolaryngol. 2007 Jan;71(1):1-6. doi: 10.1016/j.ijporl.2006.08.009. Epub 2006 Sep 25. PMID 16997385
- [Background] Bonuck KA, Freeman K, Henderson J. Growth and growth biomarker changes after adenotonsillectomy: systematic review and meta-analysis. Arch Dis Child. 2009 Feb;94(2):83-91. doi: 10.1136/adc.2008.141192. Epub 2008 Aug 6. PMID 18684748
- [Background] Wijga AH, Scholtens S, Wieringa MH, Kerkhof M, Gerritsen J, Brunekreef B, Smit HA. Adenotonsillectomy and the development of overweight. Pediatrics. 2009 Apr;123(4):1095-101. doi: 10.1542/peds.2008-1502. PMID 19336367
- [Background] Villa MP, Paolino MC, Castaldo R, Vanacore N, Rizzoli A, Miano S, Del Pozzo M, Montesano M. Sleep clinical record: an aid to rapid and accurate diagnosis of paediatric sleep disordered breathing. Eur Respir J. 2013 Jun;41(6):1355-61. doi: 10.1183/09031936.00215411. Epub 2012 Sep 27. PMID 23018902
- [Background] Chervin RD, Hedger K, Dillon JE, Pituch KJ. Pediatric sleep questionnaire (PSQ): validity and reliability of scales for sleep-disordered breathing, snoring, sleepiness, and behavioral problems. Sleep Med. 2000 Feb 1;1(1):21-32. doi: 10.1016/s1389-9457(99)00009-x. PMID 10733617
- [Background] Melendres MC, Lutz JM, Rubin ED, Marcus CL. Daytime sleepiness and hyperactivity in children with suspected sleep-disordered breathing. Pediatrics. 2004 Sep;114(3):768-75. doi: 10.1542/peds.2004-0730. PMID 15342852
- [Background] Alexopoulos EI, Kostadima E, Pagonari I, Zintzaras E, Gourgoulianis K, Kaditis AG. Association between primary nocturnal enuresis and habitual snoring in children. Urology. 2006 Aug;68(2):406-9. doi: 10.1016/j.urology.2006.02.021. PMID 16904463
- [Background] Franco RA Jr, Rosenfeld RM, Rao M. First place--resident clinical science award 1999. Quality of life for children with obstructive sleep apnea. Otolaryngol Head Neck Surg. 2000 Jul;123(1 Pt 1):9-16. doi: 10.1067/mhn.2000.105254. PMID 10889473
- [Background] Constantin E, McGregor CD, Cote V, Brouillette RT. Pulse rate and pulse rate variability decrease after adenotonsillectomy for obstructive sleep apnea. Pediatr Pulmonol. 2008 May;43(5):498-504. doi: 10.1002/ppul.20811. PMID 18383115
- [Background] Brodsky L. Modern assessment of tonsils and adenoids. Pediatr Clin North Am. 1989 Dec;36(6):1551-69. doi: 10.1016/s0031-3955(16)36806-7. PMID 2685730
- [Derived] Papadakis CE, Chaidas K, Chimona TS, Zisoglou M, Ladias A, Proimos EK, Miligkos M, Kaditis AG. Assessing the need for adenotonsillectomy for sleep-disordered breathing in a community setting: A secondary outcome measures analysis of a randomized controlled study. Pediatr Pulmonol. 2019 Oct;54(10):1527-1533. doi: 10.1002/ppul.24427. Epub 2019 Jul 3. PMID 31270970
- [Derived] Papadakis CE, Chaidas K, Chimona TS, Asimakopoulou P, Ladias A, Proimos EK, Miligkos M, Kaditis AG. Use of Oximetry to Determine Need for Adenotonsillectomy for Sleep-Disordered Breathing. Pediatrics. 2018 Sep;142(3):e20173382. doi: 10.1542/peds.2017-3382. Epub 2018 Aug 7. PMID 30087199

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment between June 2013 and April 2016; ENT Clinic of a Regional Hospital in Greece (Chania, Crete).
Groups:
- AT (Adenotonsillectomy) Group: Group underwent AT (adenotonsillectomy) immediately after the baseline nocturnal oximetry evaluation
  Adenotonsillectomy (AT): Standard surgical intervention for treatment of Obstructive SDB.
- Control Group: No AT (adenotonsillectomy) for 3 months after the baseline nocturnal oximetry evaluation.
Period: Overall Study
Arm/Group | AT (Adenotonsillectomy) Group | Control Group
Started | 93 | 93
Completed | 68 | 72
Not Completed | 25 | 21
Not completed — Baseline oximetry not acceptable | 11 | 7
Not completed — Follow-up oximetry not acceptable | 10 | 7
Not completed — Lost to Follow-up | 4 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | AT (Adenotonsillectomy) Group | Control Group | Total
Number analyzed (Participants) | 68 | 72 | 140
Age, Continuous [Mean (Standard Deviation); unit: years] | 5.9 (1.6) | 6 (1.6) | 6 (1.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 34 | 67
  Male | 35 | 38 | 73
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Greece | 68 | 72 | 140
Tonsillar size 3+ [Count of Participants; unit: Participants] — Brodsky score Upon inspection of the oropharynx
  grade 1 indicates that the tonsils are hidden in the pillars grade 2 indicates that the tonsils are beyond the anterior pillar and occupy between 25 and 50% of the pharyngeal space grade 3 indicates that the tonsils are beyond the pillars but not to the middle and occupy >50% and up to 75% of the pharyngeal space grade 4 indicates that the tonsils occupy >75% of the pharyngeal space
  Participants | 61 | 65 | 126
Tonsillar size 4+ [Count of Participants; unit: Participants] | 7 | 7 | 14
Body mass index z-score [Mean (Standard Deviation); unit: units on a scale] — The Z-score indicates the number of standard deviations away from the mean. A Z-score of 0 is equal to the mean of a reference population (i.e., healthy, age and sex-matched). Negative numbers indicate values lower than the reference population and positive numbers indicate values higher than the reference population,
  units on a scale | 0.3 (1.4) | 0.2 (1.6) | 0.2 (1.5)
Obese [Count of Participants; unit: Participants] | 12 | 14 | 26
Overweight or obese [Count of Participants; unit: Participants] | 25 | 28 | 53
Failure to thrive [Count of Participants; unit: Participants] — Body mass index (BMI) z-score <-1.645
  The Z-score indicates the number of standard deviations away from the mean. A Z-score of 0 is equal to the mean of a reference population (i.e., healthy, age and sex-matched). Negative numbers indicate values lower than the reference population and positive numbers indicate values higher than the reference population,
  Participants | 6 | 12 | 18
OSA-18 total score [Mean (Standard Deviation); unit: units on a scale] — OSA-18 questionnaire is a disease-specific QOL instrument for pediatric OSA. Caregivers are inquired in five domains (18 questions): sleep disturbance, physical symptoms, emotional symptoms, daytime function, and caregiver concerns. A score ranging from one to seven is assigned to each OSA-18 item, in which ''1'' corresponds to ''never'' and ''7'' to ''always''. OSA-18 values range from 18 to 126. Higher score corresponds to worse quality of life.
  units on a scale | 59.4 (16.3) | 58.3 (15.7) | 58.8 (15.9)

OUTCOME MEASURES:

1. Primary Outcome: Change in Number of Subjects Without Oxygenation Abnormalities
Description: Change in number of participants with a McGill oximetry score =1 (usual oxygen saturation of hemoglobin-SpO2>95%; fewer than 3 drops below 90%; and fewer than 3 clusters of desaturation events) between 3 months and 0 months.
  McGill oximetry score=1: normal or inconclusive nocturnal oximetry; McGill oximetry score=2: mild hypoxemia; McGill oximetry score=3: moderate hypoxemia; McGill oximetry score=4: severe hypoxemia.
Time Frame: 3 months (follow-up), 0 months (baseline)
Population: Subjects with a McGill oximetry score =1 or with a McGill oximetry score >1
Measure: Count of Participants; unit: Participants
Arm/Group | AT (Adenotonsillectomy) Group | Control Group
Number analyzed (Participants) | 68 | 72
Participants | 12 | 10
Statistical Analysis 1: Comparison: AT (Adenotonsillectomy) Group vs Control Group; Test type: Superiority; p = 0.54, Chi-squared; Odds Ratio (OR) = 1.3, 95% CI 2-sided [0.5 to 3.3]

2. Primary Outcome: Change in Number of Subjects Without Oxygenation Abnormalities
Description: Number of subjects who achieved a desaturation index (≥3% drop) of <2 episodes/h at 3 months (follow-up), if they had a desaturation index of ≥ 3.5 episodes/h at 0 months (baseline)
Time Frame: 3 months (follow-up), 0 months (baseline)
Population: Subjects with a desaturation index of ≥ 3.5 episodes/h at 0 months (baseline)
Measure: Count of Participants; unit: Participants
Arm/Group | AT (Adenotonsillectomy) Group | Control Group
Number analyzed (Participants) | 32 | 38
Participants | 14 | 2
Statistical Analysis 1: Comparison: AT (Adenotonsillectomy) Group vs Control Group; Test type: Superiority; p < 0.001, Chi-squared; Odds Ratio (OR) = 14, 95% CI 2-sided [2.9 to 68.4]

3. Secondary Outcome: Symptoms Predicting Obstructive Sleep Apnea (OSA)
Description: Change in Pediatric Sleep Questionnaire sleep-related breathing disorder (PSQ-SRBD) scale, between follow-up and baseline.
  PSQ-SRBD scale ranges between 0 and 1. PSQ-SRBD score <0.33 is associated with low risk of apnea-hypopnea index >5 episodes/h; PSQ-SRBD score >=0.33 is associated with high risk of apnea-hypopnea index >5 episodes/h.
Time Frame: 3 months (follow-up), 0 months (baseline)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | AT (Adenotonsillectomy) Group | Control Group
Number analyzed (Participants) | 68 | 72
score on a scale | -0.32 (0.15) | -0.01 (0.09)
Statistical Analysis 1: Comparison: AT (Adenotonsillectomy) Group vs Control Group; Test type: Superiority; p < 0.001, t-test, 2 sided; Mean Difference (Net) = -0.31, 95% CI 2-sided [-0.35 to -0.27]

4. Secondary Outcome: Quality of Life (OSA-18 Score)
Description: Change in obstructive sleep apnea (OSA)-18 total score between follow-up and baseline.
  OSA-18 is a quality of life survey including 18 questions on sleep disturbance, physical symptoms, emotional symptoms, daytime function and caregiver concerns. It is used to assess the impact of obstructive sleep apnea on child's life. Scores less than 60 suggest a small impact, between 60 and 80 moderate impact and above 80 a large impact. OSA-18 score ranges between 18 and 126.
Time Frame: 3 months (follow-up), 0 months (baseline)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | AT (Adenotonsillectomy) Group | Control Group
Number analyzed (Participants) | 68 | 72
score on a scale | -32.4 (16.9) | -0.8 (9.1)
Statistical Analysis 1: Comparison: AT (Adenotonsillectomy) Group vs Control Group; Test type: Superiority; p < 0.001, t-test, 2 sided

5. Secondary Outcome: Sleepiness
Description: Change in Modified Epworth Sleepiness Scale between follow-up and baseline
  Modified Epworth Sleepiness Scale ranges from 0 to 24; higher score indicates more daytime sleepiness.
Time Frame: 3 months (follow-up), 0 months (baseline)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | AT (Adenotonsillectomy) Group | Control Group
Number analyzed (Participants) | 68 | 72
score on a scale | -2.75 (3.07) | 0.01 (2.04)
Statistical Analysis 1: Comparison: AT (Adenotonsillectomy) Group vs Control Group; Test type: Superiority; p < 0.001, t-test, 2 sided; Mean Difference (Net) = -2.76, 95% CI 2-sided [-3.63 to -1.90]

6. Secondary Outcome: Somatic Growth-1
Description: Percent of subjects achieving an increase in weight z-score of at least 0.5. The Z-score indicates the number of standard deviations away from the mean. A Z-score of 0 is equal to the mean of a reference population (i.e., healthy, age and sex-matched). Negative numbers indicate values lower than the reference population and positive numbers indicate values higher than the reference population.
Time Frame: 0 months (baseline), 3 months (follow-up)
Measure: Count of Participants; unit: Participants
Arm/Group | AT (Adenotonsillectomy) Group | Control Group
Number analyzed (Participants) | 68 | 72
Participants | 23 | 21
Statistical Analysis 1: Comparison: AT (Adenotonsillectomy) Group vs Control Group; Test type: Superiority; p = 0.553, Chi-squared; Risk Ratio (RR) = 1.16, 95% CI 2-sided [0.71 to 1.89]

7. Secondary Outcome: Somatic Growth-2
Description: Percent of subjects achieving an increase in body mass index z-score of at least 0.5.
  The Z-score indicates the number of standard deviations away from the mean. A Z-score of 0 is equal to the mean of a reference population (i.e., healthy, age and sex-matched). Negative numbers indicate values lower than the reference population and positive numbers indicate values higher than the reference population,
Time Frame: 0 months (baseline), 3 months (follow-up)
Measure: Count of Participants; unit: Participants
Arm/Group | AT (Adenotonsillectomy) Group | Control Group
Number analyzed (Participants) | 68 | 72
Participants | 22 | 13
Statistical Analysis 1: Comparison: AT (Adenotonsillectomy) Group vs Control Group; Test type: Superiority; p = 0.057, Chi-squared; Risk Ratio (RR) = 1.79, 95% CI 2-sided [0.98 to 3.27]

8. Secondary Outcome: Enuresis
Description: Percent of subjects who achieved frequency of nocturnal enuresis < 1 night per week at follow-up (3 months), if they had incontinence at least 1 night per week at baseline (0 months).
Time Frame: 3 months (follow-up), 0 months (baseline)
Population: 24 of 68 participants in the AT group and 22 of 72 participants in the control group had nocturnal enuresis at baseline.
Measure: Count of Participants; unit: Participants
Arm/Group | AT (Adenotonsillectomy) Group | Control Group
Number analyzed (Participants) | 24 | 22
Participants | 10 | 4
Statistical Analysis 1: Comparison: AT (Adenotonsillectomy) Group vs Control Group; Test type: Superiority; p = 0.084, Chi-squared; Risk Ratio (RR) = 2.29, 95% CI 2-sided [0.84 to 6.25]

9. Secondary Outcome: Cardiovascular Effects-1
Description: Change in mean pulse rate between follow-up and baseline.
Time Frame: 3 months (follow-up), 0 months (baseline)
Measure: Median (Inter-Quartile Range); unit: beats per minute
Arm/Group | AT (Adenotonsillectomy) Group | Control Group
Number analyzed (Participants) | 68 | 72
beats per minute | -0.1 [-6.3 to 5.2] | -0.9 [-4.9 to 2.7]
Statistical Analysis 1: Comparison: AT (Adenotonsillectomy) Group vs Control Group; Test type: Superiority; p = 0.547, Wilcoxon (Mann-Whitney)

10. Secondary Outcome: Cardiovascular Effects-2
Description: Change in mean frequency of pulse rate rises (at least 6 beats per min) between follow-up and baseline.
Time Frame: 3 months (follow-up), 0 months (baseline)
Measure: Median (Inter-Quartile Range); unit: pulse rate rises per hour
Arm/Group | AT (Adenotonsillectomy) Group | Control Group
Number analyzed (Participants) | 68 | 72
pulse rate rises per hour | -1.2 [-7.6 to 1.1] | -0.1 [-4.6 to 3.8]
Statistical Analysis 1: Comparison: AT (Adenotonsillectomy) Group vs Control Group; Test type: Superiority; p = 0.062, Wilcoxon (Mann-Whitney)

11. Secondary Outcome: Cardiovascular Effects-3
Description: Change in morning systolic blood pressure z-score between follow-up and baseline.
  The Z-score indicates the number of standard deviations away from the mean. A Z-score of 0 is equal to the mean of a reference population (i.e., healthy, age and sex-matched). Negative numbers indicate values lower than the reference population and positive numbers indicate values higher than the reference population,
Time Frame: 3 months (follow-up), 0 months (baseline)
Measure: Median (Inter-Quartile Range); unit: z score
Arm/Group | AT (Adenotonsillectomy) Group | Control Group
Number analyzed (Participants) | 68 | 72
z score | 0.5 [-8 to 10.8] | -2 [-22 to 13]
Statistical Analysis 1: Comparison: AT (Adenotonsillectomy) Group vs Control Group; Test type: Superiority; p = 0.208, Wilcoxon (Mann-Whitney)

12. Secondary Outcome: Cardiovascular Effects-4
Description: Change in morning diastolic blood pressure z-score between follow-up and baseline.
  The Z-score indicates the number of standard deviations away from the mean. A Z-score of 0 is equal to the mean of a reference population (i.e., healthy, age and sex-matched). Negative numbers indicate values lower than the reference population and positive numbers indicate values higher than the reference population,
Time Frame: 3 months (follow-up), 0 months (baseline)
Measure: Median (Inter-Quartile Range); unit: z score
Arm/Group | AT (Adenotonsillectomy) Group | Control Group
Number analyzed (Participants) | 68 | 72
z score | -1 [-22.3 to 14.5] | -6 [-22 to 13]
Statistical Analysis 1: Comparison: AT (Adenotonsillectomy) Group vs Control Group; Test type: Superiority; p = 0.585, Wilcoxon (Mann-Whitney)

13. Secondary Outcome: Systemic Inflammation
Description: Change in morning serum C-reactive protein concentration between follow-up and baseline.
Time Frame: 3 months (follow-up), 0 months (baseline)
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | AT (Adenotonsillectomy) Group | Control Group
Number analyzed (Participants) | 68 | 72
mg/dL | 0 [0 to 0.07] | 0 [-0.17 to 0.07]
Statistical Analysis 1: Comparison: AT (Adenotonsillectomy) Group vs Control Group; Test type: Superiority; p = 0.074, Wilcoxon (Mann-Whitney)

14. Secondary Outcome: Improvement in Baseline SpO2
Description: Proportion of subjects who had an increase from baseline in SpO2 of >1.6%
Time Frame: 3 months (follow-up), 0 months (baseline)
Measure: Count of Participants; unit: Participants
Arm/Group | AT (Adenotonsillectomy) Group | Control Group
Number analyzed (Participants) | 68 | 72
Participants | 6 | 7

15. Secondary Outcome: Behavioral Abnormalities-1
Description: Change in the DuPaul Questionnaire for Parents score between follow-up and baseline.
Time Frame: 3 months (follow-up), 0 months (baseline)
Reporting Status: Not Posted

16. Secondary Outcome: Behavioral Abnormalities-2
Description: Change in the Achenbach Questionnaire for Parents score between follow-up and baseline.
Time Frame: 3 months (follow-up), 0 months (baseline)
Reporting Status: Not Posted

17. Secondary Outcome: Effects on Sympathetic Nervous System Activation
Description: Change in ratio of morning urine norepinephrine concentration to urine creatinine concentration between follow-up and baseline.
Time Frame: 3 months (follow-up), 0 months (baseline)
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 3 months
Groups:
- AT (Adenotonsillectomy) Group: Group underwent AT (adenotonsillectomy) immediately after the baseline nocturnal oximetry evaluation.
  Adenotonsillectomy (AT): Standard surgical intervention for treatment of Obstructive SDB.
Arm/Group | AT (Adenotonsillectomy) Group | Control Group
All-Cause Mortality (participants affected / at risk) | 0/68 | 0/72
Serious Adverse Events (participants affected / at risk) | 0/68 | 0/72
Other Adverse Events (participants affected / at risk) | 0/68 | 0/72

LIMITATIONS AND CAVEATS:
Oximetry was performed in-hospital and not at patients' homes.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No